CLINICAL TRIAL: NCT00753181
Title: Effects of Nutritional Products on Blood Glucose in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK21
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A1 (Experimental): Diabetes Meal Plan with Experimental Diabetes-Specific nutritional shake
  Interventions: Other: Nutritional Formula
- A2 (Active Comparator): Usual diet
  Interventions: Other: Usual diet
- A3 (Experimental): Diabetes Meal Plan with Experimental Diabetes-Specific Nutritional Shake, diabetes specific Cereal, and diabetes specific snack bars.
  Interventions: Other: Diabetes Meal Plan with experimental diabetes-specific nutritional shake, diabetes specific cereal, and diabetes specific snack bars.

INTERVENTIONS:
Other: Nutritional Formula — nutritional shake daily
  Arms: A1
Other: Usual diet — usual dietary habits
  Arms: A2
Other: Diabetes Meal Plan with experimental diabetes-specific nutritional shake, diabetes specific cereal, and diabetes specific snack bars. — nutritional shake, diabetes specific cereal and diabetes snack bar daily
  Arms: A3

SUMMARY:
To evaluate average daily blood glucose in subjects with type 2 diabetes following a Meal Plan including Diabetes-Specific products compared to average daily blood glucose in subjects following their usual diet.

ELIGIBILITY:
Inclusion Criteria:

1. type 2 diabetes
2. HbA1c >6.5% and <11.0%
3. male/non-pregnant, non-lactating female, at least 6 months postpartum
4. if female of childbearing potential, practicing method of birth control
5. Body Mass Index > 18.5 kg/m2 and < 43.0 kg/m2.
6. weight stable for past two months
7. if on anti-hypertensive, lipid-lowering, thyroid medication or hormone therapy, dosage constant for at least two months

Exclusion Criteria:

1. uses injected medications (e.g., insulin, exenatide) for glucose control.
2. history of diabetic ketoacidosis
3. current infection ; inpatient surgery, or corticosteroid treatment in the last 3 months or antibiotics in the last 3 weeks
4. active malignancy
5. states he/she has had a significant cardiovascular event < 12 weeks prior to study entry or history of congestive heart failure in the last 12 months.
6. end stage organ failure
7. active metabolic, hepatic, or gastrointestinal disease that may interfere with nutrient absorption, distribution, metabolism, or excretion (such as gastroparesis), excluding diabetes.
8. chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV.
9. use of herbals, dietary supplements, or medications, other than allowed medications, during past four weeks that could profoundly affect blood glucose.
10. symptomatic in response to blood collection prior to enrollment into this study.
11. clotting or bleeding disorders.
12. non-typical eating pattern
13. is currently using diabetes-specific nutritional product(s)defined as more than one eating occasion per week.
14. engages in strenuous exercise five or more times per week.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Average daily blood glucose level | 11 days

SECONDARY OUTCOMES:
Percentage of time in specified glucose ranges; Glycemic excursions; Change in plasma glucose, insulin, free fatty acids, triglycerides, 1,5-anhydroglucitol, and fructosamine; Dietary intake variables | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Vikkie Mustad, PhD, Study Director — Abbott Nutrition
Locations (2):
- United States (2):
  - Provident Clinical Research, Bloomington, Indiana
  - Radiant Research, Cincinnati, Ohio